CLINICAL TRIAL: NCT05639088
Title: Improving Transition Care for Adolescents and Young Adults With Type 1 Diabetes: A Randomized Controlled Trial of SHIFT2
Brief Title: Improving Transition Care for Adolescents and Young Adults With Type 1 Diabetes
Acronym: SHIFT2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20024552; 1K23DK131368 (NIH)
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes Management; Transition
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: SHIFT2 (Experimental): Adolescents and young adults will engage in routine medical visits and attend 6 sessions (1x/month) focused on transition preparation and diabetes management with a transition coach and will receive bi-weekly messages during these 6-months that encourage self-management behaviors.
  Parents will attend 2 sessions (month 1 and 6) with a transition coach and will receive materials, complementing their child's lesson, 1x/month for months 2-5 that focus on transition their role and supporting their child's diabetes management.
  Interventions: Behavioral: Transition preparation program
- Group B: TAU+/Control (Placebo Comparator): Participants will engage in routine medical visits and will receive education materials monthly (1x/month) regarding healthcare transition and diabetes management.
  Interventions: Other: Educational materials

INTERVENTIONS:
Behavioral: Transition preparation program — AYA will participate in virtual or in-person sessions with a transition coach and receive bi-weekly messages that encourage self-management.
  Caregivers will attend a virtual or in-person session with a transition coach.
  Other Names: SHIFT2
  Arms: Group A: SHIFT2
Other: Educational materials — AYA and caregivers will receive educational materials regarding healthcare transition and diabetes management monthly for 6 months
  Arms: Group B: TAU+/Control

SUMMARY:
The purpose of this research study is to evaluate a transition preparation program designed for adolescents and young adults (AYAs) with type 1 diabetes (T1D). This transition program will support AYAs as they prepare to transition from pediatric to adult endocrinology medical care and will also include a caregiver. Results from this study will inform clinical recommendations regarding self-management best practices for AYAs with T1D prior to transitioning to adult medical care.

DETAILED DESCRIPTION:
Investigators will recruit adolescents and young adults ages 16-22 years with T1D and a parent/guardian. Families will participate in one of two 6-month treatments: 1) SHIFT2, engaging in monthly sessions with transition coaches providing education on diabetes management and healthcare transition, or 2) Enhanced treatment (TAU+), engaging in routine medical care and receiving monthly education (no coaches).

ELIGIBILITY:
Inclusion Criteria:

AYA:

1. Type 1 Diabetes diagnosis for at least 1 year (as documented in medical record)
2. 16-22 years old
3. English speaking
4. Children's Hospital of Richmond patient (Division of Pediatric Endocrinology)
5. must have a caregiver willing to participate

Caregiver:

1. Age greater than 18 years
2. Provides care to AYA and willing to participate

Exclusion Criteria:

AYA:

1. Non-English speaking
2. Significant psychiatric, cognitive, medical or developmental conditions that would impair their ability to complete assessments and/or engage in diabetes self-care behaviors (e.g., malignancies, psychosis, intellectual disability
3. Hospitalization for depression, suicidal ideation or other psychiatric disorder within the past 12 months. Life time history of psychotic disorder
4. Medically-induced diabetes or diagnosis of diabetes other than type 1 diabetes.
5. Currently pregnant, pregnant within the past 6 months, currently breastfeeding or planning to become pregnant within the next 12 months.
6. Another member of the household (other than the participating parent) is a participant or staff member on this study.
7. Participation in another research study that may interfere with this study.
8. Previous participation in the SHIFT pilot study

Caregiver:

1. Non-English speaking
2. Significant psychiatric, cognitive, developmental conditions that would impair their ability to complete assessments and/or engage in supporting the AYA with diabetes self-care behaviors (e.g., psychosis, intellectual disability)
3. Another member of the home (not AYA) is a participant/staff member on current study
4. Participation in another research study that may interfere with current study
5. Previous participation in SHIFT pilot study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C (HbA1C) | 6 months
  HbA1C will be assessed using a standard assay from a routine blood draw or an at-home testing kit
Change in transition readiness | Baseline to 6 months
  Transition readiness will be measured using the Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) scale, which will be completed by AYAs.
Change in diabetes adherence | Baseline to 6 months
  Diabetes adherence will be assessed using the Self-Care Inventory-Revised, which will be completed by both AYA and caregivers.
Attendance at clinic visits | 6 months
  Attendance at routine clinic visits will be determined from medical records and will be assessed by the number of regularly scheduled visits attended.

SECONDARY OUTCOMES:
HbA1C | 12 months
  HbA1C will be assessed using a standard assay from a routine blood draw or an at-home testing kit.
Diabetes-related events | 12 months
  Number of diabetes-related events will be determined from medical records
Change in transition readiness | Baseline to 12 months
  Transition readiness will be measured using the Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) scale, which will be completed by AYAs.
Change in diabetes adherence | Baseline to 12 months
  Diabetes adherence will be assessed using the Self-Care Inventory-Revised, which will be completed by both AYA and caregivers.
Attendance at clinic visits | 12 months
  Attendance at routine clinic visits will be determined from medical records.
Change in diabetes support | Baseline to 12 months
  Diabetes support will be assessed using the Diabetes Social Support Questionnaire - Family Version (DDSQ-Family), which will be completed by AYAs.
Change in Diabetes Distress | Baseline to 12 months
  Diabetes distress will be assessed using the Diabetes Distress Scale (DDS) for Type 1 Diabetes (DDS), which will be completed by both AYA and caregivers. AYA will complete specific versions corresponding to age (>18 or <18) and caregivers complete their own version of the measure.
Change in Self Efficacy | Baseline to 12 months
  Self-efficacy will be measured using the Self-efficacy for Diabetes Self-Management scale (SEDSM), which will be completed by AYAs.
Change in Quality of Life | Baseline to 12 months
  Quality of life will be measured using the T1D and Life (T1DAL), which will be completed by AYA and caregiver.

OTHER OUTCOMES:
Transition Status | Baseline to 12 months
  AYAs that transition from pediatric to adult T1D care will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Caccavale, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caccavale LJ, Streisand R, LaRose JG, Wickham EP 3rd, Hilliard ME, Thornton LM, Bean MK. A clinic-based healthcare transition preparation program for adolescents and young adults with type 1 diabetes: Study protocol for the SHIFT randomized clinical trial. Contemp Clin Trials Commun. 2025 May 27;46:101500. doi: 10.1016/j.conctc.2025.101500. eCollection 2025 Aug. PMID 40529395
- [Derived] Lalji R, Koh L, Francis A, Khalid R, Guha C, Johnson DW, Wong G. Patient navigator programmes for children and adolescents with chronic diseases. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD014688. doi: 10.1002/14651858.CD014688.pub2. PMID 39382077